CLINICAL TRIAL: NCT00505336
Title: The Effect of Eplerenone and Atorvastatin on Markers of Collagen Turnover in Diastolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Professor Kenneth McDonald MD, St Vincent's University Hospital, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVUH 042
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Diastolic Heart Failure
Keywords: Diastolic heart failure; Markers of collagen turnover; Statins; Aldosterone receptor blockers
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Eplerenone; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Eplerenone
  Interventions: Drug: Eplerenone
- 3 (Active Comparator): no additional treatment
  Interventions: Other: No additional treatment
- 2 (Experimental): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Eplerenone — oral Eplerenone titrated to 50mg for duration of 12 months
  Other Names: Inspra
  Arms: 1
Other: No additional treatment — normal disease modifying therapy for heart failure i.e. ACE-I, beta blockers
  Arms: 3
Drug: Atorvastatin — oral Atorvastatin 40mg
  Other Names: Lipitor
  Arms: 2

SUMMARY:
To investigate whether the medicines eplerenone or atorvastatin have a favourable effect on diastolic heart failure.

Eplerenone is a drug that has been shown to be beneficial in Chronic Heart Failure due to pump failure. It can increase life expectancy and improve symptoms in these patients. It is not known whether or not eplerenone might be beneficial in heart failure with normal pump function (diastolic heart failure).

Atorvastatin is one of a group of cholesterol lowering medicines called statins, which have been shown to reduce cardiovascular disease in patients irrespective of whether cholesterol levels are high or normal. It is not known whether atorvastatin also reduces fibrosis of the heart which is one of the causes of diastolic heart failure.

Study hypothesis

1. To investigate the impact of aldosterone antagonism or statin therapy on markers of collagen turnover in patients with diastolic heart failure.
2. To assess the impact of aldosterone antagonism or statin therapy on markers of diastolic dysfunction and indices of clinical well being in patients with diastolic heart failure.

DETAILED DESCRIPTION:
Diastolic heart failure is a significant contributor to the heart failure syndrome. However, little work has been done on the causes of diastolic heart failure, and in contradistinction to those with systolic heart failure, little is know about the aetiology and therefore, there are few effective therapies.

It is generally believed that diastolic heart failure represents a problem with compliance and relaxation of the ventricle. One possible explanation for this is thought to be an abnormality of collagen structure in the myocardium. There are data from hypertensive populations as well as from hypertensive experimental models indicating an abnormal fibrotic process in patients with hypertensive heart disease. However, there are a few data on this potential aetiological explanation for diastolic heart failure.

It is now possible to measure serum markers of fibrosis in circulating blood. Work in this area has established the reproducibility and reliability of measurements of pro-collagen I and pro-collagen III amino-terminal, secreted as the collagen molecules are released from the fibroblast. These markers have been analysed in several settings, including normal individuals, hypertensive populations and in those with established heart failure due to systolic dysfunction. Recently we have completed a study on analysis of these factors in patients with proven diastolic heart failure. These data have demonstrated an increased activity of the amino terminal pro-collagen III (PIIINP) with a trend towards an increase in the amino-terminal pro-collagen I (PINP). Other relevant markers of the fibrotic process were not altered, including metalloproteinase enzymes (MMP) and tissue inhibitors of metalloproteinase enzymes (TIMP)

These observational data support the hypothesis that diastolic heart failure may be the result of an aggressive uncontrolled myocardial fibrotic process. The purpose of this project is to assess whether aldosterone inhibition or statin therapy may have an impact on increased levels of collagen markers, and thereby have a positive influence on parameters of diastolic function. Aldosterone is known to be a potent stimulus of the fibrotic process and therefore is a likely contributor. Support for this hypothesis comes from the observation in the systolic heart failure population where the administration of an aldosterone antagonist was found to be of benefit especially in those individuals who had serum evidence of heightened fibrotic activity. Statin therapy has been shown to reduce myocardial fibrosis in a rat model. Furthermore, preliminary data presented from the EPHESUS study has shown that greater benefits of eplerenone in those receiving concomitant statin therapy. We therefore propose to analyse the impact of atorvastatin therapy or aldosterone inhibition on markers of collagen turnover and also indices of diastolic function and markers of clinical well being.

We therefore propose to analyse the impact of aldosterone inhibition or statin therapy on markers of collagen turnover and also indices of diastolic function and markers of clinical well being.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diastolic heart failure.
* Diastolic heart failure is defined as symptoms of heart failure with an ejection fraction >45%, BNP >100pg/ml and Doppler evidence of diastolic dysfunction.

Exclusion Criteria:

* Clinically unstable as defined by any change in diuretic dose in the month prior to enrolment.
* Evidence of significant inflammatory disease or hepatic disease or metabolic bone disease which may alter parameters of collagen metabolism.
* Patients already receiving statin, aldosterone or eplerenone therapy
* Pregnant women and women of child bearing age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To investigate the impact of aldosterone antagonism or statin therapy on markers of collagen turnover in patients with diastolic heart failure. | 12 months

SECONDARY OUTCOMES:
To assess the impact of aldosterone antagonism or statin therapy on markers of diastolic dysfunction by echocardiography | 12 months
To assess the impact of aldosterone antagonism or statin therapy on indices of clinical well being | 12 months
The assess the impact of aldosterone antagonism or statin therapy on diastolic indices by cardiac MRI | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ken McDonald, MD FRCP, Study Director — Heart Failure Unit, St Vincent's University Hospital; George Mak, MB MRCPI, Principal Investigator — St Vincent's University Hospital, Ireland; Niamh Murphy, MD MRCPI, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincent's University Hospital, Ballsbridge, Dublin, Ireland

REFERENCES:
- [Derived] Mak GJ, Ledwidge MT, Watson CJ, Phelan DM, Dawkins IR, Murphy NF, Patle AK, Baugh JA, McDonald KM. Natural history of markers of collagen turnover in patients with early diastolic dysfunction and impact of eplerenone. J Am Coll Cardiol. 2009 Oct 27;54(18):1674-82. doi: 10.1016/j.jacc.2009.08.021. PMID 19850207